# A dose-response study examining the contribution of GLP-1 receptor signaling to Glucagon-stimulated insulin secretion

Adrian Vella

26th March 2020

IRB# 20-003995

NCT04459338

### **Abstract**

Glucagon is an important insulin secretagogue<sup>1,2</sup> in the concentrations found within the islet<sup>3</sup>.  $\alpha$ -cell dysfunction as occurs in T2DM<sup>4,5</sup>, in prediabetes<sup>6,7</sup> or in response to FFA elevation<sup>23</sup> results in increased glucagon concentrations. In these conditions glucagon signals through the GLP-1 receptor (GLP1R) present on  $\beta$ -cells<sup>8</sup> but its net contribution to insulin secretion is unknown. In this experiment we will determine the contribution of GLP-1R signaling to glucagon-induced insulin secretion *in vivo*. To do so, we will use a dose-response experiment for glucagon-stimulated insulin secretion. The experimental conditions will then examine how glucagon-stimulated insulin secretion is modified by blockade of GLP1R blockade using exendin-9,39. This approach will complement other experiments using a glucagon bolus known to stimulate  $\beta$ -cell function<sup>21,22</sup> in the presence and absence of GLP1R blockade.

## I. <u>Hypothesis and Specific Aims</u>

Glucagon within the islet can signal the  $\beta$ -cell through GLP1R, and acts as an insulin secretagogue<sup>3,8</sup>. This signaling is blocked by exendin-9,39<sup>9,10</sup>. The relative importance of glucagon signaling through its cognate receptor or through GLP1R is unknown. Despite the lower affinity of GLP1R for glucagon<sup>11</sup>, intra-islet concentrations of glucagon are sufficiently high to stimulate GLP1R<sup>3</sup>. The other situation where this may occur is in response to pharmacologic doses of glucagon as used for  $\beta$ -cell function testing<sup>1,2</sup> or raising peripheral glucagon concentrations above fasting values<sup>5,12,13</sup>. The experiments proposed will characterize the role of GLP1R in glucagon's actions on the  $\beta$ -cell and the potential therapeutic role of dual (GLP-1R and glucagon receptor<sup>11</sup>) agonists for the treatment of T2DM and obesity. The experiments will also provide an opportunity to test glucagon's actions on insulin secretion, independently of glucose concentrations.

We will therefore address the following specific aim: -

**Specific Aim:** Determine the contribution of *GLP1R* to glucagon-stimulated insulin secretion.

1° Hypothesis: Glucagon-stimulated insulin secretion is decreased by GLP1R blockade with exendin-9,39

**2° Hypotheses:** The contribution of GLP1R to glucagon-stimulated insulin secretion is more significant at higher glucagon concentrations

### II. Background and Significance

Diabetes mellitus causes morbidity, mortality and costs in excess of ~\$170 billion/year<sup>14</sup>. The discovery of gutderived proglucagon peptides, most specifically GLP-1<sup>15</sup>, has fueled therapeutic innovations for T2DM<sup>16</sup>. Proglucagon is transcribed and translated from the glucagon gene (*GCG*) but its final fate depends on concomitant expression of prohormone-convertase (PC) enzymes<sup>17</sup>. PC-1/3 is expressed in intestinal L-cells resulting in production of GLP-1. On the other hand, PC-2 is expressed in α-cells so that glucagon is the main derivative of proglucagon produced by these cells. However, PC-1/3 expression is inducible, suggesting that extra-intestinal synthesis and secretion of GLP-1 is possible<sup>18</sup>. IL-6<sup>19</sup>, hyperglycemia<sup>20</sup> and FFA<sup>21</sup> seem to increase PC-1/3 expression in islets. **This raises the possibility that pancreatic production of GLP-1 modulates islet function in response to glucolipotoxicity and other metabolic stressors<sup>9</sup>**.

In pharmacologic concentrations, GLP-1 is a powerful insulin secretagogue. It also inhibits glucagon secretion  $^{22}$ , delays gastrointestinal transit and decreases appetite  $^{23}$ . Endogenous concentrations of active GLP-1 are much lower and transient  $^{24}$ , partly due to the ubiquity of DPP-4. Considerable GLP-1 degradation occurs close to its site of production  $^{25}$  resulting in a circulating  $T_{1/2} \sim 1 \text{min}^{26}$ . This may explain why inhibition of GLP-1 actions at GLP1R using a competitive antagonist (exendin-9,39) has little effect on postprandial glucose metabolism  $^{27,28}$ . Indeed, only one study to date has shown a post-prandial effect of exendin-9,39 in healthy humans  $^{29}$  and this can be explained by increased gastric volume prior to meal ingestion  $^{30,31}$ . On the other hand, after bariatric surgery when endogenous GLP-1 concentrations are raised several-fold, inhibition of GLP-1 action impairs insulin secretion and raises glucose concentrations slightly, but significantly  $^{28}$ .

However, the implication that endogenous GLP-1 is of little relevance outside of bariatric surgery, is at odds with the conservation of the GLP-1 sequence across vertebrates<sup>15</sup>. GLP-1 may also contribute to the 'incretin effect' – the potentiation of post-prandial insulin secretion by gut (as opposed to I.V.) nutrient delivery. Salehi et al. reported that endogenous GLP-1 enhances postprandial insulin secretion<sup>32</sup>. However, the experiment

utilized a hyperglycemic clamp as opposed to the transient meal (or meal-like) challenges in our experiments (**Fig.1**)<sup>28,33</sup>. More germane to this proposal, they also observed an effect of GLP1R blockade on insulin secretion in response to intravenous glucose alone<sup>32</sup>.



**Figure 1:** Effect of GLP-1 receptor blockade using exendin-9,39. At time 0, subjects received an intravenous glucose challenge. Exendin-9,39 raised post-challenge glucose concentrations (also fasting in T2DM). In people without diabetes, β-cell function (**A**) is impaired but this is not apparent (**B**) in people with T2DM. On the other hand, in non-diabetic subjects there is no effect on glucagon (**C**) whereas in T2DM, glucagon is increased during fasting and the first 50 minutes after the glucose challenge (**D**). \* p < 0.05. Non diabetic data from Sathananthan, M., et al. (2013) *Diabetes* 62(8): 2752-2756

Infusion of exendin-9.39 to GLP1R during an intravenous glucose challenge (that mimics the systemic appearance of a meal) impairs β-cell function in non-diabetic humans with little effect on glucagon secretion (Fig.1a,c)<sup>33</sup>. Similar effects observed in cadaveric islets from people without T2DM (Fig.2). Conversely, in people with T2DM (Fig.1b,d) or in islets isolated from diabetic humans (Fig.5), there is no effect of exendin-9.39 on βcell function, perhaps due to the degree of  $\beta$ -cell dysfunction. However, in T2DM, exendin-9,39 raises fasting glucagon and impairs its suppression by intravenous alucose in vivo (Fig.4). Our preliminary data also suggests that GLP-1 contributes to islet function outside the postprandial period; the effects differ in T2DM compared to non-diabetic subjects (Fig.1).

Although the source of fasting GLP-1 secretion is uncertain, complementary experiments in isolated human islets (and the literature<sup>9,19,34,35</sup>) strongly suggest an islet source for GLP-1 (**Fig.2**). O'Malley et al. have suggested

that islet GLP-1 expression increases with the development of diabetes<sup>36</sup>. It is also notable that exposure of islets to FFA and hyperglycemia also increases GLP-1<sup>18,37,38</sup>. Our published<sup>33</sup> and unpublished (**Fig.1**) preliminary data, as well as genetic data<sup>39</sup> shows that GLP-1 signaling through its cognate receptor in the fasting state (or during an intravenous glucose challenge) plays a role in islet function. **Understanding the physiologic role of GLP-1 secretion independently of oral intake in humans will allow us to better modulate this pathway and prevent / treat islet dysfunction in prediabetes and T2DM.** 

The other consideration is that glucagon within the islet can signal the  $\beta$ -cell through GLP1R, and acts as an insulin secretagogue<sup>3,8</sup>. This signaling is blocked by exendin-9,39<sup>9,10</sup>. The relative importance of glucagon signaling through its cognate receptor or through GLP1R is unknown. Despite the lower affinity of GLP1R for glucagon<sup>11</sup>, intra-islet concentrations of glucagon are sufficiently high to stimulate GLP1R<sup>3</sup>. The other situation where this may occur is in response to pharmacologic doses of glucagon as used for  $\beta$ -cell function testing<sup>1,2</sup> or raising peripheral glucagon concentrations above fasting values<sup>5,12,13</sup>. The experiments proposed will characterize the role of GLP1R in glucagon's actions on the  $\beta$ -cell and the potential therapeutic role of dual (GLP-1R and glucagon receptor<sup>11</sup>) agonists for the treatment of T2DM and obesity.

Glucagon dysregulation is likely to be an earlier contributor to the pathogenesis of T2DM than has been appreciated  $^{40}$ . More significantly, although I.V. administration of glucagon is used as a test of  $\beta$ -cell function  $^2$ , its role as an insulin secretagogue within the islet has been overlooked  $^3$ . Glucagon can signal the  $\beta$ -cell through GLP1R in addition to the glucagon receptor  $^8$  (and its action blocked by exendin-9,39) $^{10}$ . What role does this play in physiology and in T2DM? The experiments proposed will quantify the effects of exendin-9,39 on glucagon-stimulated insulin secretion. Complementary experiments will also explore whether glucagon-stimulated insulin secretion is altered by rs3765467, by T2DM and by acute FFA elevation to mimic metabolic stress.

#### **III. Preliminary Data**



**Figure 2**: Acute GLP1R blockade with Ex-9,39 in isolated human cadaveric islets (obtained from Prodo labs) from non-diabetic subjects (ND) decreased insulin secretion in response to hyperglycemia. This was not apparent in T2DM. Glucose-stimulated insulin secretion was assessed by static incubation of islets at low (4mM) and high (16mM) glucose ± 100nM Ex-9,39. Insulin Stimulation Index represents fold change in insulin secretion at 16/4 mM glucose. \*p<0.05 (n=3 technical repeats).

We<sup>27,28</sup> and others<sup>41,43</sup> have shown that GLP-1 in the postprandial period has little effect on post-prandial insulin secretion outside of RYGB. Intriguingly, a variant in GLP1R that increases response to GLP-1<sup>44</sup> has been shown to decrease risk of T2DM and lower fasting glucose<sup>39,45</sup>. Also, DPP-4i which raise postprandial concentrations of active GLP-1<sup>46</sup> also lower fasting glucose concentrations, suggesting that fasting GLP-1 secretion alters islet function. The literature<sup>9,19,34,35</sup> and our preliminary data (**Fig.1,2**), suggest a pancreatic source for GLP-1.

T2DM, inflammation and metabolic stress increase islet expression of GLP-1<sup>19</sup>, perhaps as an adaptive function to preserve  $\alpha$ - and  $\beta$ -cell function. Blockade of GLP1R with exendin-9,39 seems to have divergent effects in people with and without T2DM (**Fig.4,7**), perhaps because of the degree of  $\beta$ -cell dysfunction present (**Fig.4,5**). In **Specific Aim 2** (**Fig.9**) we will characterize differences (in people with and without T2DM) in islet function during fasting and hyperglycemic conditions attributable to endogenous GLP-1. We will also alter fasting FFA concentrations<sup>40</sup> to examine the role of GLP-1 during metabolic stress in people without T2DM.

Glucagon is a known insulin secretagogue<sup>1,2</sup>. Within islets, glucagon can act on the  $\beta$ -cell through GLP1R in addition to its cognate receptor<sup>3,10</sup>. The experiments will provide an opportunity to characterize the GLP1R contribution to glucagon-stimulated

insulin secretion using a range of glucagon infusion rates.

## IV. Research Design and Methods



**Study Subjects:** After approval from the Mayo Institutional Review Board, we will recruit 20 weight-stable, otherwise healthy subjects between the ages of 18-65, usina local advertising and other methods employed previously<sup>40</sup>. Subjects will have no history of active disease or diabetes. Individuals who have expressed interest participating in research will also be contacted and invited to participate the in study. Screening Visit: After overnight fast of 8 hours. subjects will present to the Clinical Research Trials Unit (CRTU) at approximately 0700. Subjects will provide written, informed consent. To ensure they are otherwise healthy.

subjects will undergo a history and limited physical examination; blood collection for complete blood count, fasting glucose, HbA<sub>1c</sub>, sodium, potassium, creatinine and urine collection to exclude pregnancy. An ECG will also be performed. The Minnesota Leisure-Time Physical Activity questionnaire will be used to assess habitual activity levels<sup>47</sup>. **Body Composition:** After informed written consent is obtained, body composition will be measured at the screening visit using dual-energy X-ray absorptiometry (iDXA scanner; GE, Wauwatosa, WI). All subjects will be instructed to follow a weight-maintenance diet (55% carbohydrate, 30% fat and 15%

protein) for at least 3 days prior to each study. **Screening OGTT:** At approximately 0900 subjects will ingest 75g glucose. Arterialized venous blood will be sampled over 2 hrs<sup>48</sup>. Glucose values at 0 and 120 minutes will be used to categorize glucose tolerance status. Subjects who have had a DEXA or OGTT in the last 3 months as part of the Vella Lab research studies or another Mayo research group, and weight is stable (+) or (-) 5 pounds, will not be retested and previously obtained values will be used.

We will study 20 subjects a total of 2 times at least a week apart in random order. All subjects will be admitted to the Mayo Clinic CRTU at 1700 hours the evening before the study. Women who could become pregnant will have a urine collection for point of care pregnancy testing. Following ingestion of a standard 10 kcal/kg caffeine-free meal, subjects will fast overnight. The following morning at approximately 0530 (-210 min), a dorsal hand vein will be cannulated and placed in a heated Plexiglas box maintained at 55°C to allow sampling of arterialized venous blood. The contralateral forearm vein will be cannulated for glucose, and hormone infusions. At approximately 0600 (-180 min), a primed, (10μCi prime, 0.1μCi/min continuous) infusion containing trace amounts of glucose labeled with [3-3H] glucose will be started and continued till 0900 (0 min). Subsequently, the infusion will be varied so as to mimic the anticipated pattern of fall of EGP to minimize changes in Specific Activity<sup>49</sup>. At that time another glucose infusion, also labeled with [3-3H] glucose will commence and infusion rate varied so as to produce peripheral glucose concentrations of ~160mg/dL. A glucagon infusion at 0.4ng/Kg/min will start at 0900 (0 min), increasing by 0.2ng/kg/min every hour (Fig.3). Blood will be sampled till the end of the study (1400 - 300 min) when I.V. cannulas will be removed; participants will consume a late lunch and leave the CRTU. This will be referred to as the saline (Sal) day because 0.9% Saline will be infused between 0 and 300 min. On another study day, exendin-9,39 (Exe) will be infused at 300pmol/kg/min between 0 and 300 min.

**Analytical Techniques:** All blood will be immediately placed on ice, centrifuged at 4°C, separated and stored at -80°C until assay. *Glucose* will be measured using a Yellow Springs glucose analyzer. *Glucagon* will be collected in protease inhibitor-containing tubes (BD800, BD Franklin Lakes, NJ) and measured using an ELISA (Mercodia, Winston-Salem, NC). *C-peptide* will be measured using EMD Millipore (Billerica, MA) reagents. *Insulin* will be measured using a chemiluminescence assay with reagents obtained from Beckman (Access Assay, Beckman, Chaska, MN). *Total and Intact GLP-1* will be collected in protease inhibitor-containing tubes (BD800, BD Franklin Lakes, NJ) and measured using an ELISA (ALPCO Diagnostics, Salem, NH). *[3-3H] glucose specific activity* will be measured by liquid scintillation counting after deproteinization and passage over anion- and cation-exchange columns<sup>50</sup>.

**Calculations:** In addition to fasting, peak and nadir <u>hormone concentrations</u>, we will calculate area above basal (AAB) or area under the curve (AUC) during the experiment using the trapezoidal rule as previously described<sup>50</sup>. <u>S<sub>i</sub>, Insulin Secretion Rate (ISR) and β-Cell responsivity (Φ)</u> indices will be calculated<sup>51</sup> from the glucose, insulin and C-peptide concentrations observed during the experiments using the minimal model<sup>52</sup>, incorporating age-associated changes in C-peptide kinetics<sup>53</sup>. Φ is derived from the sum of  $\phi_1$  (1st phase insulin secretion) and  $\phi_2$  (2nd phase insulin secretion) as before<sup>44</sup>. Disposition index (DI) will express β-cell function as a function of the prevailing insulin action<sup>51</sup>. <u>Glucose disappearance (Rd)</u> will be calculated using steady state Steele equations<sup>54,55</sup> after <u>Specific activity</u> is smoothed as previously described<sup>56</sup>. <u>Endogenous glucose production (EGP)</u> will be calculated as the difference between the tracer determined rate of glucose appearance and the glucose infusion rate. All infusion rates will be expressed as Kg per lean body mass.

| Power Calculation | Mean ± SD | Detectable<br>difference |
|---|---|---|
| 1° hypothesis (n = 20 - paired) | | |
| Φ (10 <sup>-9</sup> min <sup>-1</sup> ) - hyperglycemia | 149 ± 45 | 30 (20%) |
| <b>Table 1:</b> Means ± SD used to estimate power | | |

**Statistical Analysis:** A paired 2-tailed student *t*-test (parametric) or a Wilcoxon rank-sign test (non-parametric) will be used to examine differences between **Sal** and **Exe** days for the 1° hypothesis (**Table 3**).

3) Power Calculation: Please refer to Table 3.

3) Interpretation: If glucagon stimulates insulin secretion by acting, at least partially, through GLP1R we would expect that exendin-9,39 will decrease the response to glucagon by blocking GLP1R. To test our 1° hypothesis, we will compare  $\Phi$  during each glucagon infusion rate in the presence and absence of exendin-9,39. Assuming that glucagon concentrations as encountered in the islet are necessary to stimulate insulin secretion via GLP1R, we expect differences to be more marked at the higher glucagon infusion rates (2° hypothesis). The experiments will be conducted in relatively lean, healthy and insulin sensitive humans. Under these experimental conditions, we expect EGP to be suppressed and insulin secretion stimulated by hyperglycemia and glucagon infusion. The rising infusion rates of glucagon will enable us to examine the

| effects of the latter on endogenous glucose presence and absence of GLP1R blockade. | production | (EGP) | and | endogenous | insulin | secretion | in | the |
|---|---|---|---|---|---|---|---|---|

## **Bibliography**

- 1. Service, F.J., *et al.* The classification of diabetes by clinical and C-peptide criteria. A prospective population-based study. *Diabetes Care* **20**, 198-201 (1997).
- 2. Robertson, R.P., *et al.* Arginine is preferred to glucagon for stimulation testing of beta-cell function. *Am J Physiol Endocrinol Metab* **307**, E720-727 (2014).
- 3. Finan, B., Capozzi, M.E. & Campbell, J.E. Repositioning Glucagon Action in the Physiology and Pharmacology of Diabetes. *Diabetes* (2019).
- 4. Muller, W.A., Faloona, G.R., Aguilar-Parada, E. & Unger, R.H. Abnormal alpha-cell function in diabetes. Response to carbohydrate and protein ingestion. *N Engl J Med* **283**, 109-115 (1970).
- 5. Shah, P., Basu, A., Basu, R. & Rizza, R. Impact of lack of suppression of glucagon on glucose tolerance in humans. *Am J Physiol* **277**, E283-290 (1999).
- Sharma, A., et al. Impaired Insulin Action is Associated with Increased Glucagon Concentrations in Non-Diabetic Humans. J Clin Endocrinol Metab 103, 314-319 (2018).
- 7. Varghese, R.T., *et al.* Mechanisms Underlying the Pathogenesis of Isolated Impaired Glucose Tolerance in Humans. *J Clin Endocrinol Metab* **101**, 4816-4824 (2016).
- 8. Moens, K., et al. Dual glucagon recognition by pancreatic beta-cells via glucagon and glucagon-like peptide 1 receptors. *Diabetes* **47**, 66-72 (1998).
- 9. Song, Y., et al. Gut-Proglucagon-Derived Peptides Are Essential for Regulating Glucose Homeostasis in Mice. *Cell Metab* (2019).
- 10. Capozzi, M.E., et al. beta Cell tone is defined by proglucagon peptides through cAMP signaling. *JCI Insight* **4**(2019).
- 11. Finan, B., et al. A rationally designed monomeric peptide triagonist corrects obesity and diabetes in rodents. *Nature Medicine* **21**, 27-36 (2015).
- 12. Shah, P., et al. Lack of suppression of glucagon contributes to postprandial hyperglycemia in subjects with type 2 diabetes mellitus. *J Clin Endocrinol Metab* **85**, 4053-4059 (2000).
- 13. Cegla, J., et al. Co-infusion of low-dose glucagon-like peptide-1 (GLP-1) and glucagon in man results in a reduction in food intake. *Diabetes* (2014).
- 14. Albright, A.L. & Gregg, E.W. Preventing type 2 diabetes in communities across the U.S.: the National Diabetes Prevention Program. *American journal of preventive medicine* **44**, S346-351 (2013).
- 15. Kieffer, T.J. & Habener, J.F. The glucagon-like peptides. *Endocr Rev* 20, 876-913 (1999).
- 16. Drucker, D.J. Evolving Concepts and Translational Relevance of Enteroendocrine Cell Biology. *The Journal of clinical endocrinology and metabolism*, jc20153449 (2015).
- 17. Holst, J.J., *et al.* Proglucagon processing in porcine and human pancreas. *J Biol Chem* **269**, 18827-18833 (1994).
- 18. Kilimnik, G., Kim, A., Steiner, D.F., Friedman, T.C. & Hara, M. Intraislet production of GLP-1 by activation of prohormone convertase 1/3 in pancreatic alpha-cells in mouse models of ss-cell regeneration. *Islets* **2**, 149-155 (2010).
- 19. Ellingsgaard, H., et al. Interleukin-6 enhances insulin secretion by increasing glucagon-like peptide-1 secretion from L cells and alpha cells. *Nat Med* **17**, 1481-1489 (2011).
- 20. Marchetti, P., et al. A local glucagon-like peptide 1 (GLP-1) system in human pancreatic islets. *Diabetologia* **55**, 3262-3272 (2012).
- 21. Ellingsgaard, H., *et al.* Interleukin-6 regulates pancreatic alpha-cell mass expansion. *Proc Natl Acad Sci U S A* **105**, 13163-13168 (2008).
- 22. Nauck, M.A., *et al.* Normalization of fasting hyperglycaemia by exogenous glucagon-like peptide 1 (7-36 amide) in type 2 (non-insulin-dependent) diabetic patients. *Diabetologia* **36**, 741-744 (1993).

- 23. Vella, A. & Camilleri, M. The Gastrointestinal Tract as an Integrator of Mechanical and Hormonal Response to Nutrient Ingestion. *Diabetes* **66**, 2729-2737 (2017).
- 24. Smushkin, G., et al. Defects in GLP-1 Response to an Oral Challenge Do Not Play a Significant Role in the Pathogenesis of Prediabetes. *J Clin Endocrinol Metab* **97**, 589-598 (2012).
- 25. Hansen, L., Deacon, C.F., Orskov, C. & Holst, J.J. Glucagon-like peptide-1-(7-36)amide is transformed to glucagon-like peptide-1-(9-36)amide by dipeptidyl peptidase IV in the capillaries supplying the L cells of the porcine intestine. *Endocrinology* **140**, 5356-5363 (1999).
- 26. Vahl, T.P., Paty, B.W., Fuller, B.D., Prigeon, R.L. & D'Alessio, D.A. Effects of GLP-1-(7-36)NH2, GLP-1-(7-37), and GLP-1- (9-36)NH2 on intravenous glucose tolerance and glucose-induced insulin secretion in healthy humans. *J Clin Endocrinol Metab* **88**, 1772-1779 (2003).
- 27. Shah, M., et al. Contribution of endogenous glucagon-like peptide-1 to changes in glucose metabolism and islet function in people with type 2 diabetes four weeks after Roux-en-Y gastric bypass (RYGB). *Metabolism* **93**, 10-17 (2019).
- 28. Shah, M., *et al.* Contribution of endogenous glucagon-like peptide 1 to glucose metabolism after Roux-en-Y gastric bypass. *Diabetes* **63**, 483-493 (2014).
- 29. Deane, A.M., *et al.* Endogenous glucagon-like peptide-1 slows gastric emptying in healthy subjects, attenuating postprandial glycemia. *J Clin Endocrinol Metab* **95**, 215-221 (2010).
- 30. Delgado-Aros, S., *et al.* Effect of GLP-1 on gastric volume, emptying, maximum volume ingested, and postprandial symptoms in humans. *Am J Physiol Gastrointest Liver Physiol* **282**, G424-G431 (2002).
- 31. Delgado-Aros, S., *et al.* Effects of glucagon-like peptide-1 and feeding on gastric volumes in diabetes mellitus with cardio-vagal dysfunction. *Neurogastroenterol Motil* **15**, 435-443 (2003).
- 32. Salehi, M., Aulinger, B., Prigeon, R.L. & D'Alessio, D.A. Effect of endogenous GLP-1 on insulin secretion in type 2 diabetes. *Diabetes* **59**, 1330-1337 (2010).
- 33. Sathananthan, M., et al. Direct Effects of Exendin-(9,39) and GLP-1-(9,36) amide on Insulin Action, beta-Cell Function, and Glucose Metabolism in Nondiabetic Subjects. *Diabetes* **62**, 2752-2756 (2013).
- 34. Traub, S., *et al.* Pancreatic alpha Cell-Derived Glucagon-Related Peptides Are Required for beta Cell Adaptation and Glucose Homeostasis. *Cell Rep* **18**, 3192-3203 (2017).
- 35. Hutch, C.R., *et al.* The role of GIP and pancreatic GLP-1 in the glucoregulatory effect of DPP-4 inhibition in mice. *Diabetologia* **62**, 1928-1937 (2019).
- 36. O'Malley, T.J., Fava, G.E., Zhang, Y., Fonseca, V.A. & Wu, H. Progressive change of intra-islet GLP-1 production during diabetes development. *Diabetes/metabolism research and reviews* **30**, 661-668 (2014).
- 37. Nie, Y., et al. Regulation of pancreatic PC1 and PC2 associated with increased glucagon-like peptide 1 in diabetic rats. *J Clin Invest* **105**, 955-965 (2000).
- 38. Vasu, S., Moffett, R.C., McClenaghan, N.H. & Flatt, P.R. Responses of GLP1-secreting L-cells to cytotoxicity resemble pancreatic beta-cells but not alpha-cells. *J Mol Endocrinol* **54**, 91-104 (2015).
- 39. Kwak, S.H., et al. Nonsynonymous Variants in PAX4 and GLP1R Are Associated With Type 2 Diabetes in an East Asian Population. *Diabetes* 67, 1892-1902 (2018).
- 40. Shah, M., et al. TCF7L2 Genotype and alpha-Cell Function in Humans Without Diabetes. *Diabetes* **65**, 371-380 (2016).
- 41. Jimenez, A., Casamitjana, R., Viaplana-Masclans, J., Lacy, A. & Vidal, J. GLP-1 Action and Glucose Tolerance in Subjects With Remission of Type 2 Diabetes After Gastric Bypass Surgery. *Diabetes Care* **36**, 2062-2069 (2013).
- 42. Jimenez, A., *et al.* GLP-1 and glucose tolerance after sleeve gastrectomy in morbidly obese subjects with type 2 diabetes. *Diabetes* **63**, 3372-3377 (2014).
- 43. Jorgensen, N.B., *et al.* Exaggerated glucagon-like peptide 1 response is important for improved beta-cell function and glucose tolerance after Roux-en-Y gastric bypass in patients with type 2 diabetes. *Diabetes* **62**, 3044-3052 (2013).

- 44. Sathananthan, A., et al. Common genetic variation in GLP1R and insulin secretion in response to exogenous GLP-1 in nondiabetic subjects: a pilot study. *Diabetes Care* **33**, 2074-2076 (2010).
- 45. Suzuki, K., *et al.* Identification of 28 new susceptibility loci for type 2 diabetes in the Japanese population. *Nat Genet* **51**, 379-386 (2019).
- 46. Dalla Man, C., et al. Dipeptidyl peptidase-4 inhibition by vildagliptin and the effect on insulin secretion and action in response to meal ingestion in type 2 diabetes. *Diabetes Care* **32**, 14-18 (2009).
- 47. Taylor, H.L., *et al.* A questionnaire for the assessment of leisure time physical activities. *J Chronic Dis* **31**, 741-755 (1978).
- 48. Sathananthan, A., et al. A concerted decline in insulin secretion and action occurs across the spectrum of fasting and postchallenge glucose concentrations. Clin Endocrinol (Oxf) 76, 212-219 (2012).
- 49. Vella, A. & Rizza, R.A. Application of isotopic techniques using constant specific activity or enrichment to the study of carbohydrate metabolism. *Diabetes* **58**, 2168-2174 (2009).
- 50. Smushkin, G., et al. The effect of a bile acid sequestrant on glucose metabolism in subjects with type 2 diabetes. *Diabetes* **62**, 1094-1101 (2013).
- 51. Cobelli, C., et al. The oral minimal model method. Diabetes 63, 1203-1213 (2014).
- 52. Breda, E., Cavaghan, M.K., Toffolo, G., Polonsky, K.S. & Cobelli, C. Oral glucose tolerance test minimal model indexes of beta-cell function and insulin sensitivity. *Diabetes* **50**, 150-158 (2001).
- 53. Van Cauter, E., Mestrez, F., Sturis, J. & Polonsky, K.S. Estimation of insulin secretion rates from C-peptide levels. Comparison of individual and standard kinetic parameters for C-peptide clearance. *Diabetes* **41**, 368-377 (1992).
- 54. Steele, R., Bjerknes, C., Rathgeb, I. & Altszuler, N. Glucose uptake and production during the oral glucose tolerance test. *Diabetes* **17**, 415-421 (1968).
- 55. Steele, R., Wall, J.S., De Bodo, R.C. & Altszuler, N. Measurement of size and turnover rate of body glucose pool by the isotope dilution method. *Am J Physiol* **187**, 15-24 (1956).
- 56. Bradley, D.C., Steil, G.M. & Bergman, R.N. OOPSEG: a data smoothing program for quantitation and isolation of random measurement error. *Comput Methods Programs Biomed* **46**, 67-77 (1995).